CLINICAL TRIAL: NCT01531205
Title: Neoadjuvant Chemohormonal Therapy Followed by Salvage Surgery for High Risk PSA Failure With Biopsy Proven Local Recurrence After Initial Definitive Radiotherapy
Brief Title: Neoadjuvant Chemohormonal Therapy Followed by Salvage Surgery for High Risk PSA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16684
Record Dates: First submitted 2012-02-08; First posted 2012-02-10 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Cancer
Keywords: recurrent; high risk
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence | interventions — Goserelin; Leuprolide; bicalutamide; cabazitaxel; Salvage Therapy; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug and Hormonal Therapy with Salvage Surgery (Experimental): Androgen Ablation (hormonal therapy before surgery), Cabazitaxel (chemotherapy before surgery), Salvage Surgery (radical prostatectomy), Post-operative Hormonal Therapy, Post-operative Follow-up
  Interventions: Drug: Androgen Ablation; Drug: Cabazitaxel; Drug: Salvage Therapy; Drug: Neoadjuvant Treatment - Hormonal Therapy; Drug: Neoadjuvant Treatment - Cabazitaxel

INTERVENTIONS:
Drug: Androgen Ablation — All patients will receive luteinizing hormone-releasing hormone (LHRH) agonist therapy (leuprolide or goserelin acetate) concurrent with Cabazitaxel, before surgery. A course of bicalutamide 50 mg daily orally for 14-21 days is recommended for patients starting LHRH agonist therapy and suspected to be at risk for tumor flare, e.g., significant obstructive urinary symptoms and will be optional in other patients.
  Other Names: goserelin acetate (Zoladex®); leuprolide acetate (Lupron®); bicalutamide (Casodex®)
Drug: Cabazitaxel — Intravenous treatment with Cabazitaxel 25 mg/m^2 is given on day 1 every 21 days. A cycle of chemotherapy will be defined as 21 days. A total of four cycles of combination therapy are planned for a total duration of 12 weeks (before surgery), starting within 3 weeks of protocol entry, to be given concurrent with hormone therapy.
  Other Names: Jevtana®
Drug: Salvage Therapy — Patients will undergo 4 cycles of chemotherapy in conjunction with LHRH agonist therapy (before surgery) subsequent to which they will have their serum Prostate-specific antigen (PSA), bone scan, abdominal pelvic computed tomography (CT) or magnetic resonance imaging (MRI) repeated. Patients with a detectable metastatic diseases will be removed from the study. Salvage surgery will be performed within 8 weeks after the completion of Cabazitaxel chemotherapy. For patients who achieved undetectable PSA following surgery, androgen deprivation therapy will be discontinued.
  Other Names: prostatectomy
Drug: Neoadjuvant Treatment - Hormonal Therapy — All treatment will be given on an outpatient basis. Treatment should start within 3 weeks of protocol entry. All patients will receive androgen ablation with LHRH agonist therapy in conjunction with the 4 cycles of Cabazitaxel for neoadjuvant chemohormonal therapy. Androgen ablative therapy will be discontinued before surgery. A course of bicalutamide 50 mg daily orally for 14-21 days is recommended for patients starting LHRH agonist therapy and suspected to be at risk for tumor flare, e.g., significant obstructive urinary symptoms and will be optional in other patients.
Drug: Neoadjuvant Treatment - Cabazitaxel — All treatment will be given on an outpatient basis and should start within 3 weeks of protocol entry. Intravenous treatment with Cabazitaxel is given on Day 1 every 3 weeks. A cycle of combination therapy will be defined as 3 weeks. A total of 4 cycles of combination therapy are planned before surgery for a total duration of 12 weeks.
  Cabazitaxel will be administered before surgery by one-hourly infusions via central or peripheral intravenous access at a dose of 25 mg/m^2 as a one hour intravenous infusion in combination with oral prednisone 10 mg administered daily throughout Cabazitaxel treatment. It is advised that all patients receiving Cabazitaxel have a reliable form of venous access, e.g., central venous catheter to ensure their ability to receive therapy without undue delay.
  Other Names: Jevtana®

SUMMARY:
The aim of this study is to test whether adding chemotherapy/cabazitaxel and hormonal/androgen deprivation therapy before surgical removal of your prostate would improve the outcome of salvage surgery for locally recurrent prostate cancer after the initial primary radiation therapy.

DETAILED DESCRIPTION:
In this study, all participants will receive cabazitaxel chemotherapy, which is approved as a second line chemotherapy for treating metastatic prostate cancer. Standard hormone or androgen ablation therapy will also be used as part of the chemohormonal therapy prior to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy must be more than 10 years
* Peripheral neuropathy: must be </= grade 1
* A minimum PSA of 1 ng/ml if not on androgen deprivation therapy
* Patients must have one of the following criteria to be eligible:

  * PSA recurrence with a doubling time of less than 9 months (calculated by at least 3 PSA values that were obtained at least 4 weeks apart)
  * Prostatic biopsy Gleason Grade of >/= 8 at the time of initial biopsy prior to radiation therapy and as determined by either an outside pathology report or on review of slides by our institutional pathologist(s)
  * Clinical stage of >/= T3 (defined as evidence of extracapsular or seminal vesicle extension on digital rectal examination or transrectal ultrasonography) either at the time of initial diagnosis or following radiotherapy
* Prior radiation therapy of any type including external beam radiotherapy, brachytherapy, high dose radiotherapy, or proton therapy
* Positive prostate biopsy documenting local recurrence following radiation therapy
* Prior androgen deprivation therapy up to a total duration of 36 months is allowable.
* Patients who are on LHRH analog therapy should continue such therapy provided that the patient does not have castration resistant prostate cancer (rising PSA in the presence of castrate levels of serum testosterone, ie < 50 ng/dl). Androgen deprivation therapy other than LHRH analog should be discontinued 4 weeks prior to study enrollment.
* All prostatic carcinoma variants except small cell carcinoma of the prostate will be allowed.
* Patients must have no evidence of metastatic diseases on the bone scan and an abdominal/pelvic CT or MRI performed within 30 days of study enrollment.
* All patients must be regarded as acceptable anesthetic risk for salvage surgery (salvage radical prostatectomy, salvage cystoprostatectomy, salvage total pelvic exenteration) and confirm their intention to undergo salvage surgery at the end of the neoadjuvant chemohormonal therapy.
* Patients must have adequate bone marrow function defined as an absolute peripheral granulocyte count of > 1,500/mm^3 and platelet count of > 100,000/mm^3; adequate hepatic function defined with a total bilirubin of < 1.5 mg/dl and aspartic transaminase/alanine transaminase (AST/ALT) < 1.5 X the upper limits of normal (ULN); adequate renal function defined as serum creatinine clearance > 60 ml/min (measured or calculated).
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution.
* All patients must be evaluated in the Department of Genitourinary Oncology prior to signing informed consent.

Exclusion Criteria:

* Patients with small cell histology
* Patients with clinical, radiological, or pathological evidence of bone, lymph node or visceral metastasis (liver or lung metastasis)
* Castration resistant prostate cancer defined as rising PSA profile in setting of castrate levels of testosterone (serum testosterone < 50 ng/dl)
* Prior chemotherapy
* Patients with severe or uncontrolled intercurrent infection
* Patients with New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina or history of myocardial infarction within the last 6 months
* Contraindications to corticosteroids
* Uncontrolled severe hypertension, persistently uncontrolled diabetes mellitus, oxygen dependent lung disease, chronic liver disease or HIV infection
* Second malignancies (excluding non-melanoma skin cancer) unless disease-free for 3 years
* Overt psychosis, mental disability or otherwise incompetent to give informed consent
* Patients with a history of severe hypersensitivity reaction to Cabazitaxel® or other drugs formulated with polysorbate 80

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Pow-Sang, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Moffitt Cancer Center from May 15, 2012 to September 27, 2013.
Groups:
- Experimental: Drug and Hormonal Therapy With Salvage Surgery: Androgen Ablation (hormonal therapy before surgery), Cabazitaxel (chemotherapy before surgery), Salvage Surgery (radical prostatectomy), Post-operative Hormonal Therapy, Post-operative Follow-up
Period: Overall Study
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Started | 2
Completed | 1
Not Completed | 1
Not completed — Did not proceed to surgery | 1

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 69 [68 to 70]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Surgical Margin Negative Rate (SM Rate)
Description: Post surgery percentage of participants with negative surgical margin. To determine the surgical margin negative rate in patients who have undergone chemohormonal therapy followed by surgery for biopsy proven androgen-dependent high risk locally recurrent prostate cancer following primary radiation therapy. Margin: The edge or border of the tissue removed in cancer surgery. The margin is described as negative or clean when the pathologist finds no cancer cells at the edge of the tissue, suggesting that all of the cancer has been removed. The margin is described as positive or involved when the pathologist finds cancer cells at the edge of the tissue, suggesting that all of the cancer has not been removed.
Time Frame: One Year
Population: Participants who proceeded to surgery
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Number analyzed (Participants) | 1
percentage of participants | 100

2. Secondary Outcome: Incidence of PSA Progression Free Survival (PFS)
Description: Percentage of participants with stable (has not increased) or undetectable PSA post surgery. To assess Prostate-specific antigen(PSA)-progression free survival and prostate cancer specific survival for patients treated by chemohormonal therapy followed by salvage surgery for biopsy proven androgen-dependent high-risk locally recurrent prostate cancer following radiation therapy.
Time Frame: Four Months
Population: Participants who proceeded to surgery
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Number analyzed (Participants) | 1
percentage of participants | 0

3. Secondary Outcome: Incidence of Complete Response (CR)
Description: Percentage of participants with CR post surgery. To evaluate the pathological complete response rate to androgen ablation plus Cabazitaxel in patients with locally recurrent prostate cancer following radiation therapy. Pathological Complete Response (pCR): Participants with no residual cancer in the local resection specimen and pelvic lymph nodes will be considered pCR.
Time Frame: One Year
Population: Participants who proceeded to surgery
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Number analyzed (Participants) | 1
percentage of participants | 0

4. Secondary Outcome: Incidence of Perioperative and Postoperative Morbidity
Description: Number of events. To access the perioperative and postoperative morbidity with salvage surgery after neoadjuvant hormonal ablation and Cabazitaxel.
Time Frame: One Year
Population: Participants who proceeded to surgery
Measure: Number; unit: events
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Number analyzed (Participants) | 1
events | 0

5. Secondary Outcome: Incidence of Detecting Circulating Tumor Cells (CTC)
Description: To determine the feasibility of detecting circulating tumor cells in this patient population. CTC results per patient in milliliters.
Time Frame: One Year
Population: All participants
Measure: Number; unit: CTC/mL
Groups:
- Participant One; Participant Two: Androgen Ablation (hormonal therapy before surgery), Cabazitaxel (chemotherapy before surgery), Salvage Surgery (radical prostatectomy), Post-operative Hormonal Therapy, Post-operative Follow-up
Arm/Group | Participant One | Participant Two
Number analyzed (Participants) | 1 | 1
CTC/mL
  Baseline CTC/mL | 2 | 1
  1 Month CTC/mL | 1 | 6
  3 Month CTC/mL | 27 | NA — Participant withdrew
  Baseline CTC Clusters/mL | 1 | 0
  1 Month CTC Clusters/mL | 0 | 2
  3 Month CTC Clusters/mL | 28 | NA — Participant withdrew
  Baseline Apop/mL | 1 | 1
  1 Month Apop/mL | 1 | 4
  3 Month Apop/mL | 1 | NA — Participant withdrew
  Baseline Small Cells/mL | 0 | 0
  1 Month Small Cells/mL | 0 | 0
  3 Month Small Cells/mL | 0 | NA — Participant withdrew
  Baseline CK-CTC/mL | 3 | 0
  1 Month CK-CTC/mL | 0 | 1
  3 Month CK-CTC/mL | 18 | NA — Participant withdrew

ADVERSE EVENTS:
Time Frame: One year
Description: All participants
Arm/Group | Experimental: Drug and Hormonal Therapy With Salvage Surgery
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Drug and Hormonal Therapy With Salvage Surgery (N=2)
Fatigue (General disorders) | 2 (3)
Pain (General disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was closed early due to low accrual. Investigators had planned to follow 25 participants from On Study through End of Follow-up, up to 10 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes